CLINICAL TRIAL: NCT01132378
Title: Mini-midvastus vs. Medial Parapatellar Approach for Minimally Invasive Total Knee Arthroplasty
Brief Title: Midvastus Versus Medial Parapatellar Approach for Minimally Invasive Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heekin Orthopedic Research Institute (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Principal Investigator, R. David Heekin, R. David Heekin, M.D., Heekin Orthopedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-01-01
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2012-02

CONDITIONS: Osteoarthritis
Keywords: Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mini-midvastus approach (Active Comparator): Mini Midvastus approach with skin incision less than 13 cm long and vastus medialis obliquus dissection not more than 3 cm from the patellar margin was used to perform total knee arthroplasty in 40 patients.
  Interventions: Procedure: Total knee arthroplasty
- Medial Parapatellar Approach (Active Comparator): Mini Medial Parapatellar approach with skin incision less than 13 cm. The extension into quadriceps tendon did not exceed 3 cm.Mini medial parapatellar approach was used to perform total knee arthroplasty.
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — staged bilateral total knee arthroplasty (not more than 7 days between surgeries)
  Other Names: Stryker Triathlon posterior stabilized components

SUMMARY:
The purpose of this study is to compare two different surgical approaches for total knee replacement surgery. The mini-midvastus approach involves cutting less of the thigh muscle (quadriceps) tendon than the classic approach (median parapatellar) in order to implant the knee components. Both will have the same skin incision.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or non-pregnant female between the ages of 21-80.
2. Patient requires cemented primary total knee replacement.
3. Patient has a diagnosis of osteoarthritis (OA), traumatic arthritis (TA) or avascular necrosis (AVN).
4. Patient has intact collateral ligaments.
5. Patient has signed and dated an IRB approved study specific consent form.
6. Patient is able and willing to participate in the study according to the protocol for the full length of the expected term of follow-up, and to follow their physician's directions.
7. Patient has failed to respond to conservative treatment modalities.

Exclusion Criteria:

1. Patient has had a prior procedure of high tibial osteotomy, cruciate ligament reconstruction or patellectomy of the surgical knee.
2. Patient is morbidly obese, >60% over ideal body weight for frame and height.
3. Patient has a deformity at the involved knee greater than 45 degrees of flexion, 45 degrees of varus or 45 degrees of valgus.
4. Patient has an active or suspected latent infection in or about the knee joint.
5. Patient has a malignancy in the area of the involved knee joint.
6. Patient has a diagnosed systemic disease that would affect the subject's welfare or overall outcome of the study (i.e. moderate to severe osteoporosis, Paget's disease) or is immunologically suppressed, or receiving steroids in excess of physiologic dose requirements.
7. Patient has a neurological deficit, which interferes with the patient's ability to limit weight bearing or places an extreme load on the implant during the healing period.
8. Female patient is or plans to become pregnant during the course of the study.
9. Patient has a known sensitivity to device materials.
10. Patient has prior diagnosis of diabetic or peripheral neuropathy in operative extremity or other neurologic disease affecting limb strength
11. Patient's bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. David Heekin, M.D., Principal Investigator — Heekin Institute for Orthopedic Research
Locations (1):
- Heekin Orthopedic Specialists, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty consecutive patients who underwent staged bilateral TKA (within no more than 7 days)were assessed at 2,6, 12 weeks and 6,12, and24 months postoperatively
Pre-assignment Details: Forty consecutive patients who underwent staged bilateral Total Knee Arthroplasty were prospectively randomised to receive mini MedialParapatellar Approach in one knee and mini-midvastus approach in the other knee (left or right)within no more than 7 days.
Groups:
- Mini-midvastus Incision: Total knee arthroplasty : staged bilateral total knee arthroplasty
  Forty consecutive patients who underwent staged bilateral Total Knee Arthroplasty were prospectively randomised to receive mini-midvastus approach in one knee and mini-Medial Parapatellar Approachthe in another knee (left or right)within no more than 7 days.
Period: Overall Study
Arm/Group | Mini-midvastus Incision
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Forty consecutive patients who underwent staged bilateral Total Knee Arthroplasty were prospectively randomised to receive mini MedialParapatellar Approach in one knee and mini-midvastus approach in the other knee (left or right)within no more than 7 days.
Groups:
- Median Parepatellar Approach or Minimidvastus Approach: Total knee arthroplasty : staged bilateral total knee arthroplasty
Arm/Group | Median Parepatellar Approach or Minimidvastus Approach
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.13 (6.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Score
Description: The higher the score the better is the result (0-100). The knee society score reflects the outcomes and perception of the patients regarding function and pain
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: score
Groups:
- Medial Parapatellar Approach: Forty consecutive patients who underwent staged bilateral Total Knee Arthroplasty were prospectively randomised to receive mini MedialParapatellar Approach in one knee and mini-midvastus approach in the other knee (left or right)within no more than 7 days.
- Mini-midvastus Approach: Total knee arthroplasty : staged bilateral total knee arthroplasty
Arm/Group | Medial Parapatellar Approach | Mini-midvastus Approach
Number analyzed (Participants) | 40 | 40
score | 98.70 (2.32) | 99.03 (1.92)

2. Secondary Outcome: Quadriceps Strength
Time Frame: 2 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Midvastus or Medial Parapatellar Approach: Forty consecutive patients who underwent staged bilateral Total Knee Arthroplasty were prospectively randomised to receive mini MedialParapatellar Approach in one knee and mini-midvastus approach in the other knee (left or right)within no more than 7 days.
Arm/Group | Midvastus or Medial Parapatellar Approach
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
The strength of the study is the standardized surgical protocol performed by a single surgeon and a prospectively randomized consecutive and blinded subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No